CLINICAL TRIAL: NCT02143843
Title: An Open-Label Extension (OLE) Study to Evaluate the Safety of the ForSight VISION5 Product in Subjects With Open-Angle Glaucoma or Ocular Hypertension Who Have Completed Study FSV5-002
Brief Title: An Open-Label Extension Study to Evaluate the Safety of the ForSight VISION5 Product
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ForSight Vision5, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FSV5-003
Record Dates: First submitted 2014-05-18; First posted 2014-05-21 (Estimated); Results first posted 2019-02-26 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2019-01

CONDITIONS: Primary Open-Angle Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Bimatoprost

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 13 mg Bimatoprost Ocular Insert (Experimental): 13 mg Bimatoprost Ocular Insert used continuously for 7 months, then replaced with a new 13 mg Bimatoprost Ocular Insert and used continuously for another 6 months.
  Interventions: Drug: Bimatoprost

INTERVENTIONS:
Drug: Bimatoprost — Bimatoprost Ocular Insert used continuously for 7 months, then replaced with a new Bimatoprost Ocular Insert and used continuously for another 6 months.
  Other Names: "Lumigan" is the branded name of bimatoprost in eye drop form

SUMMARY:
This study evaluates the long-term (13-months) safety of the Bimatoprost Ocular Insert in participants with Glaucoma or Ocular Hypertension who completed study FSV5-002. All participants received Bimatoprost Ocular Insert and wore it for approximately 7 months, then had the Insert removed and a new insert placed for another 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Completed FSV5-002 study.
2. Written informed consent prior to any study procedure.
3. Willingness to comply with the visit schedule.

Exclusion Criteria:

1. Participation in an investigational drug or device study other than FSV5-002 within the past 6 months or anticipated participation during the study period.
2. Subjects who will require contact lens use during the study period.
3. Any condition or situation (such as uncontrolled systemic disease) that, in the Investigator's opinion, might confound the results of the study, may put the subject at significant risk or might interfere with the subject's ability to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2014-06-05 (Actual); Primary Completion 2015-12-31 (Actual); Study Completion 2016-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Chen, PhD, Study Director — Allergan
Locations (10):
- United States (10):
  - Sall Medical Research Center, Artesia, California
  - Scripps Clinic Torrey Pines, La Jolla, California
  - Eye Research Foundation, Newport Beach, California
  - UC Davis Dept of Ophthalmology & Vision Science, Sacramento, California
  - Coastal Research Associates, Atlanta, Georgia
  - Clayton Eye Center, Morrow, Georgia
  - Ophthalmology Consultants, St Louis, Missouri
  - UNC Kittner Eye Center, Chapel Hill, North Carolina
  - Apex Eye, Madeira, Ohio
  - Ophthalmology Associates PC, Fort Worth, Texas

REFERENCES:
- [Derived] Brandt JD, DuBiner HB, Benza R, Sall KN, Walker GA, Semba CP; Collaborators. Long-term Safety and Efficacy of a Sustained-Release Bimatoprost Ocular Ring. Ophthalmology. 2017 Oct;124(10):1565-1566. doi: 10.1016/j.ophtha.2017.04.022. Epub 2017 May 17. No abstract available. PMID 28528010

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 13 mg Bimatoprost Ocular Insert
Started | 75
Completed | 63
Not Completed | 12
Not completed — Adverse Event | 8
Not completed — Lack of Efficacy | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | 13 mg Bimatoprost Ocular Insert
Number analyzed (Participants) | 75
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.27 (9.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44
  Male | 31

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Ocular and Non-ocular Adverse Events (AE) by Severity
Description: An AE was defined as any untoward medical occurrence (eg, sign, symptom, disease, syndrome, intercurrent illness) that occurred in a study participant, regardless of the suspected cause during the study. An ocular AE is an AE that occurred in the eye and non-ocular is an AE that occurred not in the eye. The investigator assessed the worst severity of each AE as: Mild=aware of sign or symptom, but readily tolerated, Moderate=discomfort enough to cause interference with usual activity or Severe=incapacitating with inability to work or do usual activity.
Time Frame: 13 months
Population: Safety population included all randomized participants who had ocular inserts placed in their eyes.
Measure: Number; unit: percentage of participants
Arm/Group | 13 mg Bimatoprost Ocular Insert
Number analyzed (Participants) | 75
percentage of participants
  Ocular, Mild | 53.3
  Ocular, Moderate | 14.7
  Ocular, Severe | 1.3
  Non-ocular, Mild | 12.0
  Non-ocular, Moderate | 18.7
  Non-ocular, Severe | 1.3

2. Secondary Outcome: Change From Baseline in Mean Intraocular Pressure (IOP)
Description: IOP is a measurement of the fluid pressure inside the eye. Diurnal IOP measurements were taken at 8 am (Time (T)=0 hour), 10 am (T=2 hour), and 4 pm (T=8 hour) at Months 3, 6, 7 and 13. IOP readings from both eyes were averaged to compute a single IOP value for each diurnal time-point, then averaged over 0, 2, and 8 hour to get the mean IOP. The change from baseline in mean IOP was calculated. The median value over the 13 month period is reported. A negative change from Baseline indicated an improvement. Baseline is defined as the IOP assessment done at the last visit (Month 6) of study FSV5-002 [NCT01915940].
Time Frame: Baseline (Day 1) to Month 13
Population: Full Analysis Set (FAS) included all randomized participants who had ocular inserts placed in their eye and who had at least 1 on-treatment study visit completed,
Measure: Median (Inter-Quartile Range); unit: mm Hg
Arm/Group | 13 mg Bimatoprost Ocular Insert
Number analyzed (Participants) | 75
mm Hg | -4 [-6 to -2]

ADVERSE EVENTS:
Time Frame: Start of this Open-Label Extension Study to Last Visit (Up to 13 Months)
Arm/Group | 13 mg Bimatoprost Ocular Insert
Serious Adverse Events (participants affected / at risk) | 1/75
Other Adverse Events (participants affected / at risk) | 42/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 13 mg Bimatoprost Ocular Insert (N=75)
Urinary tract infection (Infections and infestations) | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 13 mg Bimatoprost Ocular Insert (N=75)
Conjunctival hyperaemia (Eye disorders) | 15
Punctate keratitis (Eye disorders) | 12
Eye discharge (Eye disorders) | 11
Vision blurred (Eye disorders) | 9
Eye pruritus (Eye disorders) | 6
Dry eye (Eye disorders) | 5
Foreign body sensation in eyes (Eye disorders) | 5
Ocular discomfort (Eye disorders) | 4
Upper respiratory tract infection (Infections and infestations) | 6
Lacrimation increased (Eye disorders) | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No presentation or publication of Institution's data relating to the Trial may occur until after the Trial has been completed at all sites. If Investigator desires to present or publish, investigator must submit any and all manuscripts, posters, abstracts, or other intended publications (hereinafter collectively referred to as "manuscripts") to Sponsor at least sixty (60) days prior to the actual submission of such manuscript(s) for publication.